CLINICAL TRIAL: NCT03211884
Title: Evidence-Based Mental Health Services for Distressed Post-9/11 Military Family Caregivers
Brief Title: Effects of PSTon Mental Health Outcomes in Caregivers of Post-9/11 Combat Veterans With a Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Chatham University (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-16-1-0690
Record Dates: First submitted 2017-06-07; First posted 2017-07-07 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Military Family; Brain Injuries, Traumatic
Keywords: Problem solving therapy; Military family caregivers; Cognitive impariment; Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trail.
Masking Description: Self-administered on-line surveys which preclude the need for a masked outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem-solving therapy (Experimental): Couched within Bandura's social-cognitive theory, self-management refers to the process by which individuals accept responsibility for and take action to change their behaviors, obtain knowledge related to their situation (e.g., behavioral manifestations of a TBI) through increased awareness and use of effective personal resources (e.g., skill in every-day problem-solving). This ultimately enhances the caregivers' confidence that they can cope with caregiving and behavior-related stressors in the care recipient.
  Interventions: Behavioral: Problem-Solving Thearpy
- Usual Care (No Intervention): Usual care was defined as various military caregiver organizations, support groups and services available to all family caregivers of combat Veterans (e.g., Military OneSource; Operation We Are Here; Veterans Administration Program of Comprehensive Assistance for Family Caregivers; American Red Cross Military and Veteran Caregiver Network; Project New Hope; Wounded Veteran Family Care; Women for Wounded Warriors).

INTERVENTIONS:
Behavioral: Problem-Solving Thearpy — The problem-solving therapy (PST)-based intervention consists of nine, 60-90 minute educational sessions conducted face-to-face via the Internet (through video conferencing software) approximately 2 weeks apart. After attending a preliminary 15 minute "meet & greet" session, participants received written and verbal education about solving everyday problems. Together, the participant and interventionist complete the 7-steps to solve at least one problem together before ending the training. Participants keep a record of their problem-solving efforts between sessions and questions they had related to the application of PST. These records were used as a basis for discussion during the PST training sessions.
  Other Names: PST
  Arms: Problem-solving therapy

SUMMARY:
The primary aim of this study is to assess the efficacy of PST for positively impacting distressed military family caregiver's depression and burden levels (secondary outcomes), ultimately enhancing their mental health quality of life (QOL, primary outcome).

DETAILED DESCRIPTION:
Background: Traumatic brain injury (TBI) is considered the "signature injury" of recent conflicts in Iraq and Afghanistan, with 22% of returning troops experiencing a TBI. After receiving acute and rehabilitative healthcare services, combat veterans with a TBI (active Service Members and Veterans) are typically cared for at home, by their female (79%) parent (62%, 32% spouses), and the majority (60%) of these caregivers receive little or no help from others with their caregiving responsibilities. Not only is TBI a well-documented risk factor for dementia of the Alzheimer's type (AD) later in life, noteworthy similarities exist between the experiences of family caregivers of Veterans with TBI and caregivers of civilians with AD. Symptoms of a TBI are very similar to AD and include cognitive impairment (deficits in memory, language, attention, and/or planning), difficulty communicating, poor impulse control, and poor emotion regulation. Both conditions necessitate adaptation to emotional and behavioral changes in the injured family member, and personality changes may result in relationship strain between the injured person and his or her family caregiver. Similar to AD, symptoms of a TBI do not lessen over time, are often perceived as burdensome, and are associated with negative mental health outcomes in their family caregivers. Similarly, both AD and TBI family caregivers report additional stressors (e.g., continuous monitoring for unpredictable behaviors and their consequences) when cohabitating with the impaired or injured family member for an extended period of time.

Objective/Hypotheses: To improve the mental health of family caregivers of post-9/11 combat veterans with a TBI, the proposed study is designed to evaluate the efficacy of an evidence-based, short-term (9, 60-mintue session), solution-focused, self- management intervention utilizing problem-solving therapy (PST) to lessen burden and depression levels, and improve the quality of life (QOL) in co-residing family caregivers of combat veterans with a TBI (military family caregivers). PST is based on the premise that real-life problem-solving plays an important role as a mediator of the relationship between stressful life events and negative mental health outcomes. When deficits in problem-solving lead to ineffective coping attempts, under high levels of stress exposure, burden and depression is likely to ensue. Building on our previous work with caregivers of civilians with mild cognitive impairment (a proposed precursor for AD) and early-stage AD, it is hypothesized that military family caregivers receiving PST training will endorse lower levels of caregiving burden and depression, and improved mental health QOL, at each follow-up assessment, than caregivers in the comparison (usual care) group.

Specific Aims: The primary aim of this study is to assess the efficacy of PST for positively impacting distressed military family caregiver's burden, and depression levels, ultimately enhancing their mental health QOL (primary outcomes). Data will also be collected to characterize physical and social stressors for these caregivers such as illness that limits the caregiver's activities, new household management and caregiving responsibilities, satisfaction with social roles and activities, lifestyle constraints, the quality of the marital relationship, perceived social support, and demographic factors. A secondary aim of the proposed study is to determine which of a series of key caregiver sociodemographic factors moderate PST- intervention efficacy for caregiving burden and mental health QOL outcomes.

Study Design: A randomized controlled trail design (intention-to-treat model) will be used to evaluate the effects of an individualized PST-based intervention on burden, mental health, and well-being outcomes in family caregivers of combat veterans with a TBI. We expect to enroll and randomize 100 family caregivers of Veterans with a TBI from the Joint Forces Explosive Ordnance Disposal (the disarming and disposal of bombs) Warrior Foundation and Boulder Crest Retreat for Wounded Warriors family caregiver websites. Caregivers assigned to the PST group will receive nine PST training sessions (each approximately 60 minutes) delivered face-to-face every two weeks (to allow time for problem solving efforts and scheduling conflicts) using study-specific webcams (part of the Study Welcome Kit). Software will be utilized that permits recording and saving of intervention sessions for review (to ensure treatment fidelity over time). Outcomes will be collected through the Internet (to enhance the study's sustainability and scalability) and measured baseline, and at 1-, 3-, 6-, and 12-mos. post-intervention.

Study Relevance: Since family caregivers constitute the largest group of adult care providers in the United States and the market value of family caregiving exceeds that spent on formal health and nursing home care, the mental health and well-being of family caregivers of Veterans with a TBI - and their subsequent ability to assist wounded Veterans at home (e.g., prevent institutionalization of injured/impaired Veterans) - is of paramount importance. If the PST-based intervention reduces burden levels and improves mental health aspects of QOL in military family caregivers, the data will be used to lay the foundation for offering PST- based mental health services for distressed family caregivers of Veterans with a TBI through the VA Program of Comprehensive Assistance for Family Caregivers.

ELIGIBILITY:
Screen positive for caregiving burden

Lives with a post-9/11 Veteran or Service Member with a combat-related traumatic brain injury

Communicates in English

No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Mental health quality of life (QOL) | Baseline, 1, 3, 6, & 12 months post-intervention
  Mental health quality of life (QOL) is measured with the mental health component of the Medical Outcomes Survey (MOS) Health Survey Short Form-12 Version 2 (SF-12v2). MOS-SF-12V2 is a multipurpose survey of health related quality of life (both physical and mental) and a practical tool for directly linking norms from large population surveys with the results from more focused RCTs. Both Mental Component Summary Scores (MCS) and Physical Component Summary Scores (PCS) were shown to have high internal consistency reliability (alpha > .80).
Change in Subjective caregiver burden | Baseline, 1, 3, 6, & 12 months post-intervention
  Caregiving burden (worry, exhaustion) is measured with the Montgomery's Subjective Burden Scale (SBS). The SBS includes a series of 13 questions to establish how the caregiver feels about caring for their family member with dementia. The SBS demonstrated sound psychometric properties in the feasibility study (Cronbach's alpha = .95) and preliminary data shows variability in responses for the target population.

SECONDARY OUTCOMES:
Change in Depression Levels | Baseline, 1, 3, 6, & 12 months post-intervention
  Depression levels are measured with the Center for epidemiological Studies - Depression Scale (CES-D, Revised) is composed of 20 items, each response corresponds to the frequency of the symptom in the preceding week, higher score indicate more severe depressive symptoms. A cutoff score of 16 or greater is indicative of individuals at high risk for clinical depression. The CES-D demonstrated high internal reliability (Cronbach's alpha = .91) in our feasibility study.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Garand, Ph.D., Principal Investigator — Duquesne University
Locations (1):
- Duquesne University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated from the study will be made widely available, while safeguarding the privacy of participants and protecting confidential and proprietary data and third-party intellectual property. In line with the Congressionally Directed Medical Research Programs (CDMRP) policy, all unique data and final research data generated will be made available to the research community and to the public at large. Along with the data, documentation will be provided about the methodology and procedures used to collect the data, details about codes, definitions of variables, variable field locations, frequencies, and any other unique background information. The PI will share data via external storage media after the requester has completed a data-sharing agreement to impose appropriate limitations on the user.
Supporting Information: ICF
Time Frame: Follow-up data was collected until August 2020. Preliminary data analysis will be available by May 2021.